CLINICAL TRIAL: NCT04502550
Title: Subcortical-cortical Network Dynamics of Anesthesia and Consciousness
Brief Title: Brain Networks and Consciousness
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Nader Pouratian, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2021-0396
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Loss of Consciousness; Parkinson Disease; Essential Tremor; Anesthesia
Keywords: general anesthesia; deep brain stimulation; basal ganglia; thalamus; sensorimotor cortex
MeSH Terms: conditions — Unconsciousness; Parkinson Disease; Essential Tremor | interventions — Propofol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (7):
- Parkinson's Disease patients with DBS, no stimulation: This cohort will serve as as the observed group, displaying basal ganglia pathology.
  A syringe pump controlled by Stanpump implementing the Eleveld Pharmacokinetics-Pharmacodynamics (PK-PD) model for propofol will be used as a targeted controlled infusion (TCI) system to achieve plasma target propofol concentrations. Target effect-site concentration of propofol will be started at 1.4 μg/mL and will be increased by 0.3 μg/mL with reassessment until endpoints are achieved.
  Experiments will be completed with DBS off.
  Interventions: Drug: Propofol
- Essential Tremor patients with DBS: This cohort will serve as a control group (no basal ganglia pathology). A syringe pump controlled by Stanpump implementing the Eleveld Pharmacokinetics-Pharmacodynamics (PK-PD) model for propofol will be used as a TCI system to achieve plasma target propofol concentrations. Target effect-site concentration of propofol will be started at 1.4 μg/mL and will be increased by 0.3 μg/mL with reassessment until endpoints are achieved.
  Experiments will be completed with DBS off.
  Interventions: Drug: Propofol
- Parkinson's Disease patients with DBS, Gpi stimulation: This cohort will serve as as the observed group, displaying basal ganglia pathology.
  A syringe pump controlled by Stanpump implementing the Eleveld Pharmacokinetics-Pharmacodynamics (PK-PD) model for propofol will be used as a targeted controlled infusion (TCI) system to achieve plasma target propofol concentrations. Target effect-site concentration of propofol will be started at 1.4 μg/mL and will be increased by 0.3 μg/mL with reassessment until endpoints are achieved.
  Participants will be stimulated at the Gpi via DBS leads during propofol induced loss of consciousness.
  Interventions: Drug: Propofol
- Parkinson's Disease patients with DBS, Gpe stimulation: This cohort will serve as as the observed group, displaying basal ganglia pathology.
  A syringe pump controlled by Stanpump implementing the Eleveld Pharmacokinetics-Pharmacodynamics (PK-PD) model for propofol will be used as a targeted controlled infusion (TCI) system to achieve plasma target propofol concentrations. Target effect-site concentration of propofol will be started at 1.4 μg/mL and will be increased by 0.3 μg/mL with reassessment until endpoints are achieved.
  Participants will be stimulated at the Gpe via DBS leads during propofol induced loss of consciousness.
  Interventions: Drug: Propofol
- Parkinson's Disease patients undergoing DBS surgery, Gpe stimulation: A syringe pump controlled by Stanpump implementing the Eleveld Pharmacokinetics-Pharmacodynamics (PK-PD) model for propofol will be used as a targeted controlled infusion (TCI) system to achieve plasma target propofol concentrations. Target effect-site concentration of propofol will be started at 1.4 μg/mL and will be increased by 0.3 μg/mL with reassessment until endpoints are achieved.
  Participants will be stimulated at the Gpe via DBS leads, and cortical activity will be recorded via ECoG during propofol induced loss of consciousness.
  Interventions: Drug: Propofol
- Parkinson's Disease patients undergoing DBS surgery, Gpi stimulation: A syringe pump controlled by Stanpump implementing the Eleveld Pharmacokinetics-Pharmacodynamics (PK-PD) model for propofol will be used as a targeted controlled infusion (TCI) system to achieve plasma target propofol concentrations. Target effect-site concentration of propofol will be started at 1.4 μg/mL and will be increased by 0.3 μg/mL with reassessment until endpoints are achieved.
  Participants will be stimulated at the Gpi via DBS leads, and cortical activity will be recorded via ECoG during propofol induced loss of consciousness.
  Interventions: Drug: Propofol
- Parkinson's Disease patients undergoing DBS surgery, no stimulation: A syringe pump controlled by Stanpump implementing the Eleveld Pharmacokinetics-Pharmacodynamics (PK-PD) model for propofol will be used as a targeted controlled infusion (TCI) system to achieve plasma target propofol concentrations. Target effect-site concentration of propofol will be started at 1.4 μg/mL and will be increased by 0.3 μg/mL with reassessment until endpoints are achieved.
  Participants will not receive any stimulation via DBS leads, and cortical activity will be recorded via ECoG during propofol induced loss of consciousness.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Target effect-site concentration of propofol will be started at 1.4 μg/mL and will be increased by 0.3 μg/mL with reassessment until endpoints are achieved.

SUMMARY:
General anesthesia (GA) is a medically induced state of unresponsiveness and unconsciousness, which millions of people experience every year. Despite its ubiquity, a clear and consistent picture of the brain circuits mediating consciousness and responsiveness has not emerged. Studies to date are limited by lack of direct recordings in human brain during medically induced anesthesia. Our overall hypothesis is that the current model of consciousness, originally proposed to model disorders and recovery of consciousness after brain injury, can be generalized to understand mechanisms of consciousness more broadly. This will be studied through three specific aims. The first is to evaluate the difference in anesthesia sensitivity in patients with and without underlying basal ganglia pathology. Second is to correlate changes in brain circuitry with induction and emergence from anesthesia. The third aim is to evaluate the effects of targeted deep brain stimulation on anesthesia induced loss and recovery of consciousness. This study focuses on experimentally studying these related brain circuits by taking advantage of pathological differences in movement disorder patient populations undergoing deep brain stimulation (DBS) surgery. DBS is a neurosurgical procedure that is used as treatment for movement disorders, such as Parkinson's disease and essential tremor, and provides a mechanism to acquire brain activity recordings in subcortical structures. This study will provide important insight by using human data to shed light on the generalizability of the current model of consciousness. The subject's surgery for DBS will be prolonged by up to 40 minutes in order to record the participant's brain activity and their responses to verbal and auditory stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to cooperate during conscious operative procedure for up to 40 minutes
* Clinical diagnosis of Parkinson's disease or essential tremor
* Preoperative MRI without evidence of cortical or subdural adhesions or vascular abnormalities

Exclusion Criteria:

* Patients with recent use (within one week) of anticoagulant or antiplatelet agent use
* Neurocognitive testing indicating amnestic cognitive deficits
* History of intolerance of propofol or medical indications to use an anesthetic other than propofol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants are Parkinson's disease and essential tremor patients undergoing revision/replacement of an implantable pulse generator for DBS, or initial DBS implantation.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Propofol dose response curve | baseline
  Serum concentration of propofol throughout targeted infusion will be correlated with the patient's response to behavioral assessments in order to predict the time course of plasma and effect site concentration of propofol, establishing differential anesthetic sensitivity profiles.
Behavioral assessment of propofol induced loss / recovery of consciousness and responsiveness | baseline
  For each experiment, three behavioral responses will be evaluated: (1) loss/recovery of spontaneous movement (i.e., loss and recovery of responsiveness) (2) loss/recovery of movement in response to stimuli (separately to clicks [non-salient] and verbal stimuli [salient]), and (3) loss/recovery of movement to command (verbal command with patient name with instruction to open their eyes, as proxy of loss/recovery of consciousness).
Electrocorticogram (ECoG) and pallidal Local Field Potential (LFP) recordings | baseline
  Cortical ECoG and Globus Pallidus internus / Globus Pallidus externus (GPi/GPe) LFP recordings will occur during DBS implantation surgery during both induction and emergence with target-controlled infusion of propofol changes in network parameters. Neurophysiological signals will be correlated the evolution of behavioral measures of loss of consciousness and responsiveness during propofol infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Nader Pouratian, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Nader Pouratian, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No